CLINICAL TRIAL: NCT05172596
Title: A Phase 2 Study of PHE885, B-cell Maturation Antigen (BCMA)- Directed CAR-T Cells in Adult Participants With Relapsed and Refractory Multiple Myeloma.
Brief Title: PHE885 CAR-T Therapy in Adult Participants With Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated since the sponsor made the decision to discontinue further development of the study drug durcabtagene autoleucel (PHE885).
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPHE885B12201; 2021-003747-22 (EudraCT Number)
Record Dates: First submitted 2021-12-22; First posted 2021-12-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; B-cell maturation antigen; BCMA; BCMA-directed; chimeric antigen receptor; CAR-T; PHE885
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PHE885 (Experimental): Patients will receive PHE885
  Interventions: Biological: PHE885

INTERVENTIONS:
Biological: PHE885 — Intravenous (IV) infusion

SUMMARY:
This is a Phase II study to determine the efficacy and safety of PHE885, a BCMA-directed CAR-T cell therapy, manufactured with a new process. The CAR-T cell therapy will be investigated as a single agent in relapsed and refractory multiple myeloma

DETAILED DESCRIPTION:
This clinical trial employs an open label, single arm, multi-center design with primary analysis testing overall response rate ( ORR), including one interim analysis for futility and one interim analysis for efficacy.

The trial population includes adult patients with relapsed and refractory multiple myeloma (MM) after failure of 3 or more lines of therapy, including failing an immunomodulatory drug (IMiD), a proteasome inhibitor (PI) and an anti-CD38 (cluster of differentiation 38) monoclonal antibody (mAb) and who have measurable disease at enrollment per IMWG criteria . In addition, patients must be refractory to the last line of therapy

The trial will enroll 90 efficacy evaluable adult patients with relapsed and refractory MM (efficacy evaluable means participants infused with a PHE885 product at target dose 10e6 that met all release specifications).

Patients will be followed for acute and intermediate safety and efficacy within this trial for a minimum of 2 years before being transferred to the long-term follow-up trial. A long-term post-study follow-up for lentiviral vector safety will be offered under a separate destination protocol for 15 years post injection per health authority guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of informed consent form (ICF) signature
2. Adult patients after failure of three or more lines of therapy including an IMiD (e.g., lenalidomide or pomalidomide), a proteasome inhibitor (e.g., bortezomib, carfilzomib), and an approved anti-CD38 antibody (e.g., daratumumab, isatuximab), and who have documented evidence of disease progression (IMWG criteria) 3, Must have received ≥2 consecutive cycles of treatment for at least three prior regimens unless deemed refractory to that regimen (i.e., progressive disease as the best response)

4. Must be refractory to the last treatment regimen (defined as progressive disease on or within 60 days measured from last dose of last regimen).

5. Measurable disease at enrollment as defined by the protocol 6. Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening 7. Must have a leukapheresis material of non-mobilized cells accepted for manufacturing

Exclusion Criteria:

1.Prior administration of a genetically modified cellular product including prior BCMA CAR-T therapy. 2.Participants who have received prior BCMA -directed bi-specific antibodies or anti-BCMA antibody drug conjugate.

3. Prior autologous SCT within 3 month or allogenic SCT within 6 months prior to signing informed consent.

4.Plasma cell (PC) leukemia and other plasmacytoid disorders, other than MM 5.POEMS syndrome 6.Active central nervous system (CNS) involvement by malignancy 7.Patients with active neurological autoimmune or inflammatory disorders 8.Inadequate cardiac, renal, hepatic or hematologic function as defined in the protocol.

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) per Independent Review Committee (IRC) in Efficacy Analysis Set | 24 Months
  Percentage of patients with best overall response (BOR) of either stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR) according to the International Myeloma Working Group (IMWG) criteria'

SECONDARY OUTCOMES:
Key Secondary End point: MRD Negativity rate in Bone Marrow | 24 months
  Evaluate the efficacy of PHE885 with respect to MRD negativity rate in bone marrow measured by next generation sequencing (NGS)
Complete response rate (CRR) | 24 Months
  Percentage of patients with BOR of sCR or CR according to the IMWG criteria
Time to response | 24 Months
  Time form PHE885 infusion to the date of first documented response (PR or better)
Duration of Response (DOR) | 24 Months
  Time from first documented response (PR or better) until relapse or death due to any cause
Progression free survival (PFS) | 24 Months
  Time from PHE885 infusion until progression or death due to any cause
Time to next anti-myeloma treatment (TTNT) | 24 Months
  Time from PHE885 infusion until start of new anti-myeloma therapy or death due to any cause
Overall Survival (OS) | 24 Months
  Time from PHE885 infusion until death due to any cause
Durability of Minimal Residual Disease (MRD)negativity | 24 Months
  Time from the start of undetectable MRD to the time of reappearance of detectable MRD
Patient Reported Outcomes (PRO): EQ-5D-5L Health Questionnaire | 24 months
  PROs as measured by EuroQoL Group EQ-5D-5L Health Questionnaire is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.
Patient Reported Outcomes (PRO): EORTC-QLQ-C30 | 24 months
  PROs as measured by European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC-QLQ-C30) Questionnaire will be used as a measure of health-related quality of life.
Patient Reported Outcomes (PRO): EORTC-QLQ-MY20 | 24 months
  PROs as measured by EORTC-QLQ-MY20 is a 20-item myeloma module intended for use among patients varying in disease stage and treatment modality.
PHE885 manufacturing success rate | 24 Months
  Percentage of enrolled patients for whom PHE885 product was manufactured that met all release specifications
Manufacturing turnaround time | 24 months
  Time from pick of cryopreserved material at the clinic or hospital until return to the clinical or hospital
Transgene of PHE885 concentrations over time in peripheral blood and bone marrow | 24 Months
  As determined by quantitative polymerase chain reaction (qPCR)
Cellular kinetics parameter: Cmax | 24 Months
  The maximum transgene level at Tmax
Cellular kinetics parameter: Tmax | 24 Months
  The time to peak transgene level
Cellular kinetics parameter: AUC | 24 months
  The Area under the curve of the transgene level
Immunogenicity to PHE885 | 24 Months
  Summary of pre-existing and treatment-induced immunogenicity (cellular and humoral) of PHE885

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (6):
  - Stanford University, Palo Alto, California
  - Emory University School of Medicine-Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health Sciences University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fred Hutch Cancer Research, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Brazil (2):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Calgary, Alberta, Canada
- France (4):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
- Germany (4):
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Salamanca
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The Trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com